CLINICAL TRIAL: NCT07154537
Title: Immunogenicity and Safety of Pneumococcal Conjugated Vaccine 13 (PCV13) in Patients With Multiple Myeloma
Brief Title: Pneumococcal Conjugated Vaccine 13 (PCV13) for Patients With Multiple Myeloma (MM)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201511041MIND; MOHW109-TDU-B-211-114002 (Other: Ministry of Health and Welfare, Executive Yuan, Taiwan); MOHW108-TDU-B-211-133002 (Other: Ministry of Health and Welfare, Executive Yuan, Taiwan); MOHW106-CDC-C-11400104 (Other: Ministry of Health and Welfare, Executive Yuan, Taiwan)
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Immunogenicity; pneumococcal conjugated vaccine 13 (PCV13); safety
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-dose PCV13 (Experimental): 2 doses PCV13 with one month apart
  Interventions: Biological: 2-dose PCV13
- 1-dose PCV13 (Active Comparator): 1 dose PCV13
  Interventions: Biological: 1-dose PCV13

INTERVENTIONS:
Biological: 2-dose PCV13 — 2 doses PCV13 with one month apart
  Arms: 2-dose PCV13
Biological: 1-dose PCV13 — 1 dose PCV13
  Arms: 1-dose PCV13

SUMMARY:
Multiple myeloma patients often get serious infections that can be deadly. A British study looked at newly diagnosed patients and found that bacterial infections were the main cause of death in the first 60 days, mostly from pneumonia (66%) and blood poisoning (23%). The most common bacteria causing these infections were pneumococcus, staph, and E. coli.

Medical experts recommend that multiple myeloma patients get pneumonia vaccines. However, some studies show these vaccines don't work well in these patients, raising questions about whether they're really helpful. It's also unclear if patients need one shot or multiple shots like other high-risk patients.

This study at National Taiwan University Hospital will randomly give multiple myeloma patients either one or two doses of the 13-valent pneumonia vaccine. Researchers will check if the vaccine is safe and if it helps the immune system fight infections, while trying to figure out what makes the vaccine work better in some patients than others.

DETAILED DESCRIPTION:
Infection has always been a common and potentially life-threatening problem for multiple myeloma patients. A British study on newly diagnosed multiple myeloma patients investigated the causes of death within 60 days of enrollment and found that bacterial infection was the most common cause of death, followed by kidney failure, myocardial infarction, or stroke. Among patients who died from bacterial infections, 66% died from pneumonia, 23% from sepsis, and 11% from other infections. Among bacterial infection patients with culture results, Streptococcus pneumoniae was the most common pathogen, followed by Staphylococcus aureus and Escherichia coli.

The International Myeloma Working Group recommends that multiple myeloma patients receive pneumococcal vaccination. Some research findings have shown that pneumococcal vaccination in multiple myeloma patients is ineffective or very limited in effectiveness, questioning the recommendation for routine pneumococcal vaccination. Furthermore, it remains unknown whether multiple doses of vaccine are needed, as in hematopoietic stem cell transplant patients.

Therefore, for multiple myeloma patients at National Taiwan University Hospital, this study aims to randomly assign patients to receive either one or two doses of 13-valent pneumococcal conjugate vaccine, evaluate its safety and immune response generation, and identify factors related to vaccine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma
* Stable clinical condition to have vaccination at outpatient clinic

Exclusion Criteria:

* Those who have received pneumococcal vaccine within the past five years
* Unable to communicate verbally with the subject
* Subject has an active infection
* Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity to serotype 6B, 14, 23F, 19F | before every dose of PCV13, and 4 weeks, every 12 weeks for one year, and every year for 5 years after the last dose of PCV13

SECONDARY OUTCOMES:
Safety of PCV13 | within one week after each dose of PCV13
  adverse effects within one week after each dose of PCV13
invasive pneumococcal diseases | after the last dose of PCV13 for 5 years
Mortality | after the last dose of PCV13 for 5 years
  death and causes of death
Pneumonia | after the last dose of PCV13 for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Yun Sun, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan